CLINICAL TRIAL: NCT01901068
Title: A Multicentre, International, Prospective Post-market Clinical Follow-up to Evaluate MonoMax for Abdominal Wall Closure
Brief Title: MonoMax for Abdominal Wall Closure
Acronym: MULTIMAC
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1010
Record Dates: First submitted 2013-07-05; First posted 2013-07-17 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Wall Wound
Keywords: Laparotomy; Surgical Procedures, Elective; Sutures; Abdominal Wound Closure Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MonoMax: Elective primary laparotomy
  Interventions: Device: MonoMax

INTERVENTIONS:
Device: MonoMax — Abdominal wall will be closed with MonoMax after an elective primary laparotomy.

SUMMARY:
A great number of different suture techniques and suture materials are in use in order to reconstitute the abdominal wall integrity, but there is no surgical gold standard for abdominal wall closure until today. Various Meta-Analyses and randomized controlled trials have been performed, which compared non-absorbable or long-term absorbable versus rapid absorbable suture materials or monofilament versus multifilament suture materials, or continuous versus interrupted suture techniques respectively. This lack of evidence has the following outcome: burst abdomen is observed in 1-3% of patients within the first days after a laparotomy. The incidence of abdominal wall hernias 12 months postoperatively is estimated to be up to 20% (range 9 to 20%) . Wound infections develop in 3 to 21% of patients undergoing a median laparotomy within the first 30 days. At present most surgeons favour monofilament long-absorbable continuous sutures as the most suitable material for closing abdominal wounds after midline laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Elective primary laparotomy
* Written informed consent

Exclusion Criteria:

* Peritonitis
* Emergency surgery
* Severe psychiatric and neurologic disease
* Drug- and / or alcohol abuse according to local standard
* Lack of informed consent
* Current immunosuppressive therapy
* Chemotherapy within the 2 weeks before operation
* Radiotherapy of the abdomen completed less than 8 before surgery
* Pregnant or breast-feeding women
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of reoperation due to burst abdomen | participants will be followed for the duration of hospital stay, an expected average of 10 days
Frequency of wound infections | participants will be followed for the duration of hospital stay, an expected average of 10 days

SECONDARY OUTCOMES:
Incidence of wound healing until day of discharge | participants will be followed for the duration of hospital stay, an expected average of 10 days
Length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (2):
  - Chirurgicka klinika, Fakultni nemocnine, Hradec Králové
  - Chirurgicka klinika, Fakultni nemocnine, Olomouc
- Central Emergency Military Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fink C, Baumann P, Wente MN, Knebel P, Bruckner T, Ulrich A, Werner J, Buchler MW, Diener MK. Incisional hernia rate 3 years after midline laparotomy. Br J Surg. 2014 Jan;101(2):51-4. doi: 10.1002/bjs.9364. Epub 2013 Nov 26. PMID 24281948
- [Background] Fischer L, Baumann P, Husing J, Seidlmayer C, Albertsmeier M, Franck A, Luntz S, Seiler CM, Knaebel HP. A historically controlled, single-arm, multi-centre, prospective trial to evaluate the safety and efficacy of MonoMax suture material for abdominal wall closure after primary midline laparotomy. ISSAAC-Trial [NCT005725079]. BMC Surg. 2008 Jul 21;8:12. doi: 10.1186/1471-2482-8-12. PMID 18644124
- [Background] Albertsmeier M, Seiler CM, Fischer L, Baumann P, Husing J, Seidlmayer C, Franck A, Jauch KW, Knaebel HP, Buchler MW. Evaluation of the safety and efficacy of MonoMax(R) suture material for abdominal wall closure after primary midline laparotomy-a controlled prospective multicentre trial: ISSAAC [NCT005725079]. Langenbecks Arch Surg. 2012 Mar;397(3):363-71. doi: 10.1007/s00423-011-0884-6. Epub 2011 Dec 20. PMID 22183105